CLINICAL TRIAL: NCT04713059
Title: The Affiliated Hospital of Qingdao University
Brief Title: Toripalimab Combined With Anlotinib for Patients With Advanced, Relapsed, or Refractory Gastric, or Esophagogastric Junction Cancer (EGJC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhangxiaochun, The Affiliated Hospital of Qingdao University, The Affiliated Hospital of Qingdao University
Other Study IDs: CAANGC/EJGC
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Gastric or Gastro-oesophageal Junction Carcinoma; Advanced, Relapsed Gastric or Gastro-oesophageal Junction Carcinoma; Second-line Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with CPS ≥ 1 or MSI-H or TMB ≥ 10Mb/MUT
  Interventions: Genetic: FGFR2
- patients with CPS =0 , MSS and TMB < 10Mb/mut
  Interventions: Genetic: FGFR2

INTERVENTIONS:
Genetic: FGFR2 — Mutation of FGFR2

SUMMARY:
Patients were aged >18 years with histological confirmed GC/EGJC and were refractory to the first line of therapy. Additional eligibility requirements included: ≥1 measurable disease at baseline per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v 1.1); Eastern Cooperative Oncology Group Performance status of 0 or 1; or life expectancy of ≥ 3 months and adequate organ function. The main exclusion criteria were interstitial lung disease, pulmonary fibrosis, active or prior autoimmune disease or active hepatitis, or history of anlotinib or any other PD-L1/PD-1 antagonist treatment. Patients with abdominal fistula, diverticulitis, gastrointestinal ulcerative disease or perforation, or abdominal abscess within the prior 4 weeks were also excluded. This study was an open, exploratory single-arm, phase II trial. Enrolled patients received anlotinib (12mg, po. qd, d1-14) combined with toripalimab (240 mg, inv, over 30 min once every 2 weeks).

ELIGIBILITY:
Inclusion Criteria:

Patients were aged >18 years with histological confirmed GC/EGJC and were refractory to the first line of therapy. Additional eligibility requirements included: ≥1 measurable disease at baseline per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST v 1.1); Eastern Cooperative Oncology Group Performance status of 0 or 1; or life expectancy of ≥ 3 months and adequate organ function.

Exclusion Criteria:

The main exclusion criteria were interstitial lung disease, pulmonary fibrosis, active or prior autoimmune disease or active hepatitis, or history of anlotinib or any other PD-L1/PD-1 antagonist treatment. Patients with abdominal fistula, diverticulitis, gastrointestinal ulcerative disease or perforation, or abdominal abscess within the prior 4 weeks were also excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were aged >18 years with histological confirmed GC/EGJC and were refractory to the first line of therapy.
Sampling Method: Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 01.01.2019 to 01.01.2021
6m-PFS | 01.01.2019 to 01.01.2021
safety | 01.01.2019 to 01.01.2021

SECONDARY OUTCOMES:
PFS | 01.01.2019 to 01.01.2021
OS | 01.01.2019 to 01.01.2021

CONTACTS AND LOCATIONS:
Locations (1):
- Xiaochun Zhang, Qingdao, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang M, Zhang C, Hu Y, Li T, Yang G, Wang G, Zhu J, Shao C, Hou H, Zhou N, Liu K, Zhang X. Anlotinib Combined with Toripalimab as Second-Line Therapy for Advanced, Relapsed Gastric or Gastroesophageal Junction Carcinoma. Oncologist. 2022 Nov 3;27(11):e856-e869. doi: 10.1093/oncolo/oyac136. PMID 35857405